CLINICAL TRIAL: NCT04425252
Title: The CRISIS Study: A Randomized Open-label Study Assessing the Safety and Anti-coronavirus Response of Suppression of Host Nucleotide Synthesis in Hospitalized Adults With Coronavirus-19 (COVID-19)
Brief Title: Safety and Anti-coronavirus Response of Suppression of Host Nucleotide Synthesis in Patients With COVID-19
Acronym: CRISIS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clear Creek Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCB-CRISIS-01
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Results first posted 2022-02-16 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
Keywords: DHODH inhibition; antiviral; coronavirus; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — brequinar; Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized 1:2 to standard of care (SOC) alone or SOC + brequinar
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Other): Subjects are hospitalized for COVID-19 and will receive all supportive/interventional care per institutional guidelines.
  Interventions: Other: Standard of Care
- Brequinar (Experimental): Subjects will receive standard of care plus brequinar 100 mg daily (Study Days 1-5).
  Interventions: Drug: Brequinar

INTERVENTIONS:
Drug: Brequinar — DHODH inhibitor, 100 mg daily x 5 days
  Other Names: Standard of Care + Brequinar
  Arms: Brequinar
Other: Standard of Care — Standard of Care per institutional guidelines for COVID-19 patients
  Arms: Standard of Care

SUMMARY:
This will be a phase 1a randomized, open label, multi-center study with approximately 24 subjects. All subjects will receive standard of care (SOC) per institutional guidelines for treatment of hospitalized patients with COVID-19 infection. In addition to SOC, the brequinar group will receive 5 daily doses of brequinar 100 mg.

DETAILED DESCRIPTION:
This will be a phase 1a randomized, open label, multi-center study with approximately 24 subjects. All subjects will receive standard of care (SOC) per institutional guidelines for SARS-CoV-2 infection. Subjects will be randomly assigned in a 1:2 ratio to SOC alone or SOC plus brequinar. The SOC plus brequinar group will receive 5 daily doses of brequinar 100 mg on Days 1 - 5 in addition to SOC. Physical examinations, vital signs, laboratory assessments, SARS-CoV-2 testing, and other observations will be conducted by experienced personnel throughout the study based on the Schedule of Events. Blood chemistry tests include blood urea nitrogen (BUN), creatinine, alkaline phosphatase (ALP), alanine amino transferase (ALT), aspartate amino transferase (AST), bilirubin, total protein, albumin, glucose, serum electrolytes (sodium, potassium, chloride, carbon dioxide/bicarbonate, and calcium), lactate dehydrogenase (LDH). Plasma will be collected for inflammatory markers such as D-dimer, ferritin, c-reactive protein (CRP), and erythrocyte sedimentation rate (ESR). Pro-inflammatory markers will be measured. Serum is to be collected for research purposes. Hematology tests include hemoglobin, hematocrit, complete blood count with full differential, and platelet count. Nasopharyngeal swabs for viral load will be collected Days 1, 3, 5, 7, and 15. Survival will be assessed through Day 29.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent for the trial, written, electronic, verbal or other method deemed acceptable by the institution and IRB.
2. 18 years of age or older.
3. If discharged from the hospital prior to Study Day 15 or if follow up is needed for study drug-related adverse event, willing to go to an outpatient facility if feasible or be in contact with the study team (phone call or other digital media) for remaining study assessments.
4. Laboratory-confirmed SARS-CoV-2 infection as determined by real time polymerase chain reaction (RT-PCR) or other Food and Drug Administration (FDA)-cleared commercial or public health assay.
5. Hospitalized (in patient with expected duration ≥ 24 hours)
6. The effects of brequinar on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men and women treated or enrolled on this protocol must also agree to use adequate contraception for the duration of study participation and for 90 days after completion of brequinar administration.
7. Male subjects must agree to refrain from sperm donation from initial study drug administration until 90 days after the last dose of brequinar.
8. ≤ 10 days since first COVID-19 symptom as determined by treating clinician.
9. Able to swallow capsules.
10. At least one COVID-19 symptom including but not limited to fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms, shortness of breath, dyspnea, dysgeusia, or other symptom commonly associated with COVID-19.

Exclusion Criteria:

1. Any physical examination findings and/or history of any illness that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the patient.
2. Active malignancy other than squamous cell carcinoma; anticancer treatment such as chemotherapy or radiation therapy within the past month.
3. Nursing women or women of childbearing potential (WOCBP) with a positive pregnancy test.
4. Treatment with another DHODH inhibitor (e.g., leflunomide or teriflunomide), tacrolimus, sirolimus.
5. Platelets ≤150,000 cell/mm3.
6. Hemoglobin < 10 gm/dL
7. Absolute neutrophil count < 1500 cells/mm3
8. Renal dysfunction, i.e., creatinine clearance < 30 mL/min
9. AST and/or ALT > 1.5 ULN, or total bilirubin > ULN
10. History of bleeding disorders or recent surgery in the six weeks preceding enrollment
11. Concomitant use of agents known to cause bone marrow suppression leading to thrombocytopenia
12. History of gastrointestinal ulcer, or history of gastrointestinal bleeding.
13. History of hepatitis B and/or C infection, active liver disease and/or cirrhosis.
14. Heart failure, current uncontrolled cardiovascular disease, including unstable angina, uncontrolled arrhythmias, major adverse cardiac event within 6 months (e.g. stroke, myocardial infarction, hospitalization due to heart failure, or revascularization procedure).
15. Life expectancy of < 5 days in the judgment of the treating clinician.
16. Evidence of critical illness defined by at least one of the following:

    a. Respiratory failure requiring at least one of the following: i. Endotracheal intubation and mechanical ventilation, noninvasive positive pressure ventilation, ECMO, or clinical diagnosis of respiratory failure (i.e., clinical need for one of the preceding therapies, but preceding therapies may not be able to be administered in setting of resource limitation) ii. Shock (defined by systolic blood pressure < 90 mm Hg, or diastolic blood pressure < 60 mm Hg or requiring vasopressors) b. Multi-organ dysfunction/failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2021-01-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Hartford Hospital, Hartford, Connecticut
  - Baptist Medical Center, Jacksonville, Florida
  - University of South Florida/Tampa General, Tampa, Florida
  - University of New Mexico, Albuquerque, New Mexico
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Enrolled: 19 AUG 2020 Last Patient Completed the study: 12 JAN 2021 Patients were hospitalized with COVID-19 and were recruited at the hospital where they were being treated as in-patients.
Pre-assignment Details: All subjects were hospitalized as in-patients as part of the inclusion criteria. 25 patients were enrolled, but 2 withdrew consent prior to treatment and had no post-randomization assessments for a total of 23 subjects randomized in the study and included in the modified intent-to-treat population.
Groups:
- Standard of Care: Subjects were hospitalized for COVID-19 and received standard of care per institutional guidelines for COVID-19 patients.
- Standard of Care + Brequinar: Subjects were hospitalized for COVID-19 and received standard of care per institutional guidelines for COVID-19 patients plus brequinar 100 mg daily x 5 days.
Period: Overall Study
Arm/Group | Standard of Care | Standard of Care + Brequinar
Started | 8 | 15
Completed | 4 | 13
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Subject did not return due to COVID-19 restrictions. | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care: Subjects were hospitalized with COVID-19 and received institutional standard of care for COVID-19.
- Standard of Care + Brequinar: Subjects were hospitalized with COVID-19 and received institutional standard of care for COVID-19 plus brequinar 100 mg daily x 5 days.
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Standard of Care + Brequinar | Total
Number analyzed (Participants) | 8 | 15 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.38 (16.02) | 55.59 (14.78) | 54.24 (15.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 4 | 8 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 7 | 8 | 15
  More than one race | 0 | 4 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 15 | 23

OUTCOME MEASURES:

1. Primary Outcome: Safety/Tolerability Assessed by Rates of Grade 3 or 4 Post Randomization Adverse Events
Description: Safety/tolerability as assessed by number of participants with Grade 3 or 4 post randomization adverse events.
Time Frame: Through Day 15.
Population: All subjects in the Modified Intent-to-Treat Population included those with at least one post randomization assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Standard of Care + Brequinar
Number analyzed (Participants) | 8 | 15
Participants | 1 | 1

2. Primary Outcome: Safety/Tolerability as Assessed by Rates of Serious Adverse Events (SAEs).
Description: Safety/tolerability as assessed by number of participants with Serious Adverse Events (SAEs).
Time Frame: Through Day 15
Population: Modified intent-to-treat population included all subjects with at least one post randomization assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Standard of Care + Brequinar
Number analyzed (Participants) | 8 | 15
Participants | 1 | 3

3. Primary Outcome: Safety/Tolerability Measured by Mortality at Day 29
Description: Safety/tolerability as measured by mortality at Day 29
Time Frame: Through Day 29
Population: Modified intent-to-treat population included all participants with at least one post-randomization assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Standard of Care + Brequinar
Number analyzed (Participants) | 8 | 15
Participants | 0 | 0

4. Secondary Outcome: Hospitalization Status
Description: All participants were hospitalized at time of study entry. This outcome measures participant hospitalization status at Days 3, 5, 7, and 15 in terms of: hospitalized in intensive care unit (ICU), hospitalized as part of initial admission, re-hospitalized (had been discharged from initial hospitalization and was re-admitted to the hospital) or was dead at the time of the assessment.
Time Frame: Days 3, 5, 7, and 15
Population: Modified intent-to-treat population which includes all participants with at least one post-randomization study assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Standard of Care + Brequinar
Number analyzed (Participants) | 8 | 15
Participants
  Day 3 Died | 0 | 0
  Day 3 Hospitalized in ICU | 0 | 3
  Day 3 Hospitalized | 3 | 9
  Day 3 Discharged | 5 | 3
  Day 5 Died | 0 | 0
  Day 5 Hospitalized in ICU | 0 | 1
  Day 5 Hospitalized | 3 | 4
  Day 5 Discharged | 5 | 10
  Day 7 Died | 0 | 0
  Day 7 Hospitalized in ICU | 0 | 0
  Day 7 Hospitalized | 1 | 0
  Day 7 Discharged | 7 | 15
  Day 15 Died: number analyzed (Participants) | 7 | 15
  Day 15 Died | 0 | 0
  Day 15 Hospitalized in ICU: number analyzed (Participants) | 7 | 15
  Day 15 Hospitalized in ICU | 0 | 0
  Day 15 Hospitalized: number analyzed (Participants) | 7 | 15
  Day 15 Hospitalized | 1 | 1
  Day 15 Discharged: number analyzed (Participants) | 7 | 15
  Day 15 Discharged | 6 | 14
  Day 15 Missing | 1 | 0

5. Secondary Outcome: Duration of Hospitalization
Description: Duration in number of days from admission to discharge; days counted as an integer only.
Time Frame: Through Day 15
Population: The modified intent-to-treat population included all participants with at least one post-randomization assessment.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard of Care | Standard of Care + Brequinar
Number analyzed (Participants) | 8 | 15
days | 2 [1.5 to 4] | 4 [3 to 5]

6. Secondary Outcome: NEWS2 Score
Description: Measure Description: National Early Warning Score (NEWS) 2. Composite score of respiratory rate, oxygen saturation, systolic blood pressure, pulse, consciousness, and temperature. The NEWS2 provides a score of illness severity based on respiratory rate, SpO2, whether the patient is breathing room air or on oxygen, systolic blood pressure, heart rate, consciousness, and body temperature. The scale ranges from 20 (worst/sickest) to 0 (all measurements in a normal range). The NEWS2 was assessed at baseline, Days 3, 5, 7, and 15.
Time Frame: Baseline, Days 3, 5, 7, and 15.
Population: Participants with at least one post randomization assessment who were able to return to the clinic for a study visit. Multiple subjects were unable to return for scheduled study assessments at various time points due to COVID-19 restrictions in place at the institutions where the study was conducted.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Standard of Care | Standard of Care + Brequinar
Number analyzed (Participants) | 8 | 13
units on a scale
  Baseline (Day 1 pre dose) | 1.9 (0.69) | 3.9 (0.80)
  Day 3: number analyzed (Participants) | 3 | 10
  Day 3 | 3.0 (1.15) | 2.8 (0.47)
  Day 5: number analyzed (Participants) | 4 | 5
  Day 5 | 2.5 (1.55) | 3.8 (1.07)
  Day 7: number analyzed (Participants) | 4 | 4
  Day 7 | 3.3 (1.03) | 3.8 (1.75)
  Day 15: number analyzed (Participants) | 4 | 7
  Day 15 | 0.00 (0.00) | 2.6 (0.97)

ADVERSE EVENTS:
Time Frame: 29 days
Description: Events that occurred prior to informed consent were entered as medical history; AEs that occurred after informed consent were entered on the AE form. Subjects were questioned and observed for evidence of AEs, whether or not judged by the Investigator or designated person to be related to study drug.
Arm/Group | Standard of Care | Standard of Care + Brequinar
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/8 | 3/15
Other Adverse Events (participants affected / at risk) | 0/8 | 3/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=8) | Standard of Care + Brequinar (N=15)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=8) | Standard of Care + Brequinar (N=15)
Hyperglycemia (Endocrine disorders) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
CCB-CRISIS-01 was a small, open-label study with small numbers of subjects analyzed. In addition, the study was conducted prior to availability of COVID-19 vaccinations and there were many missed visits and assessments due to COVID-19 restrictions in place at the time that prohibited return visits to the hospital or clinic. Standard of care for these hospitalized subjects included remdesivir and steroids.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT04425252/Prot_002.pdf
  • Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT04425252/SAP_001.pdf